CLINICAL TRIAL: NCT04007289
Title: Apixaban for Intrahepatic Non Cirrhotic Portal Hypertension
Acronym: APIS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P170916J
Record Dates: First submitted 2019-05-24; First posted 2019-07-05 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Intrahepatic Non Cirrhotic Portal Hypertension
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Intervention Model Description: This study will be a prospective, national multicentric, phase III, superiority comparative randomized (1:1) double-blinded clinical trial with two parallel arms: apixaban versus placebo.
Who Masked: Participant
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- APIXABAN (Active Comparator): Apixaban, 1 pill of 2.5 mg per os twice a day (one in the morning and one in the evening) for 24 months.
  Interventions: Drug: Apixaban
- PLACEBO (Placebo Comparator): Placebo, 1 pill per os twice a day (one in the morning and one in the evening) for 24 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apixaban — Administration of Apixaban ; 2 clinical examinations; blood tests, 3 liver and spleen stiffness measurements, 2 contrast enhanced echocardiographies, 1 hepatic ultrasonography, Biological samples collections to identify predictors of thrombosis and liver related events
  Arms: APIXABAN
Drug: Placebo — Administration of placebo ; 2 clinical examinations; blood tests, 3 liver and spleen stiffness measurements, 2 contrast enhanced echocardiographies, 1 hepatic ultrasonography,
  Arms: PLACEBO

SUMMARY:
Intrahepatic non-cirrhotic portal hypertension (INCPH) is a rare disease mostly affecting adults in their forties, characterized by portal hypertension related to alterations of intrahepatic microcirculation in the absence of cirrhosis.The only therapeutic options currently available for patients with INCPH include prophylaxis for variceal bleeding using betablockers and/or endoscopic band ligation and TIPSS (transjugular intrahepatic portosystemic shunt) or liver transplantation for severe cases.

The investigators hypothesize that anticoagulation using Apixaban in patients with INCPH might prevent occurrence or extension of portal, splenic or mesenteric veins thromboses and thus the development of chronic portal vein thrombosis and associated complications, but also avoid intrahepatic thromboses and consequently liver disease progression and variceal bleeding.

The Primary Objective is to evaluate the effect of 24 months low dosing of apixaban (2.5 mg x 2/day) versus placebo on the occurrence or the extension of portal venous system thrombosis (including splenic, mesenteric veins, portal trunk or left or right portal branches) at 24 months in patients with INCPH.

166 patients will be included in 21 centers in a prospective, national multicentric, phase III, superiority comparative randomized (1:1) double-blinded clinical trial with two parallel arms: apixaban versus placebo.

DETAILED DESCRIPTION:
Intrahepatic non-cirrhotic portal hypertension (INCPH) is a rare disease mostly affecting adults in their forties, characterized by portal hypertension related to alterations of intrahepatic microcirculation in the absence of cirrhosis.The only therapeutic options currently available for patients with INCPH include prophylaxis for variceal bleeding using betablockers and/or endoscopic band ligation and TIPSS (transjugular intrahepatic portosystemic shunt) or liver transplantation for severe cases.

The investigators hypothesize that anticoagulation using Apixaban in patients with INCPH might prevent occurrence or extension of portal, splenic or mesenteric veins thromboses and thus the development of chronic portal vein thrombosis and associated complications, but also avoid intrahepatic thromboses and consequently liver disease progression and variceal bleeding.

The Primary Objective is to evaluate the effect of 24 months low dosing of apixaban (2.5 mg x 2/day) versus placebo on the occurrence or the extension of portal venous system thrombosis (including splenic, mesenteric veins, portal trunk or left or right portal branches) at 24 months in patients with INCPH.

The Secondary Objectives are :

1. To assess the safety of apixaban on: (a) any major bleeding as defined by the ISTH (International Society on Thrombosis and Haemostasis) guidelines; (b) liver toxicity; (c) adverse events and reactions.
2. To compare the effect of 24 months low dosing of apixaban (2.5 mg x 2/day) versus placebo on the following outcomes, assessed during the 24 months of treatment:

   1. - at least one event among: deep vein thrombosis in any location, arterial thrombosis, major bleeding, death
   2. - the occurrence of deep vein thrombosis in any location or arterial thrombosis
   3. - mortality (global, liver related, non-liver related), and mortality or liver transplantation
   4. - each and any event among: liver decompensation, complications of portal hypertension including portal hypertensive related gastrointestinal bleeding, liver transplantation or death;
   5. - portal hypertension related features (spleen size, platelet count, size of esophageal varices, portal blood flow velocity) and markers of bacterial translocation and inflammation
   6. - liver function
   7. - quality of life
3. To evaluate the effect of 24 months low dosing of apixaban (2.5 mg x 2/day) versus placebo on the occurrence or the extension of portal venous system thrombosis (including splenic, mesenteric veins, portal trunk or left or right portal branches) at 24 months after randomisation in patients with INCPH according to HIV status
4. To identify predictors of portal venous system thrombosis and liver related events:

   * in the control group: liver and spleen stiffness; portal blood flow velocity; specific coagulation tests; markers of bacterial translocation and inflammation
   * in the group receiving apixaban: plasma apixaban levels
5. To assess treatment compliance
6. To study the occurrence or extension of portal venous system thrombosis or occurrence of deep vein thrombosis in any location or arterial thrombosis in the 6 months after the 24-month treatment with apixaban versus placebo.

166 patients will be included in 21 centers in a prospective, national multicentric, phase III, superiority comparative randomized (1:1) double-blinded clinical trial with two parallel arms: apixaban versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18 and ≤ 90 year old male and female patients,
* For child-bearing aged women, contraception using progestatives, or intrauterine device or mechanical contraception
* Adequate prophylaxis against variceal bleeding according to EASL (European association for the study of the liver) guidelines
* Intrahepatic non cirrhotic portal hypertension (INCPH), defined according to the recent VALDIG workshop (Feb. 2017, Ascona, Italy) as having one of the following simultaneous associations:

  1. absence of cirrhosis on an adequate liver biopsy, and one or more signs specific for portal hypertension
  2. absence of cirrhosis on an adequate liver biopsy, and one or more signs not specific for portal hypertension and one or more histological signs for INCPH
  3. in the absence of adequate liver biopsy, 2 reliable liver stiffness values determined using transient elastography (Fibroscan) < 10 kPa and one or more signs specific for portal hypertension

Exclusion Criteria:

* Myeloproliferative disease treated with aspirin to prevent vascular events, paroxysmal nocturnal hemoglobinuria.
* Ongoing oestroprogestative contraception
* Pregnant or breastfeeding women
* Complete thrombosis of superior mesenteric vein and/or inferior mesenteric vein
* Complete portal vein thrombosis or portal cavernoma
* Recent (<6 months) partial portal venous system thrombosis
* Mandatory indication or contraindication for anticoagulation according to guidelines of the American college of chest physicians
* Concomitant treatment with any other anticoagulant agent unless when bridging from one to the other is performed
* Disease at high risk of bleeding (except for portal hypertension)
* Active clinically significant bleeding:. This may include current or recent gastrointestinal ulceration, presence of malignant neoplasms at high risk of bleeding, recent brain or spinal injury, recent brain, spinal or ophthalmic surgery, recent intracranial haemorrhage, arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities.
* Platelet < 40000/mm3, or prothrombin index <40% in the absence of anti-vitamin K or Factor V < 40% or Fibrinogen < 1.0g/L
* Transjugular intrahepatic portosystemic shunt (TIPSS) or surgical portosystemic shunt
* Participation in another interventional trial
* Creatinine clearance < 30 mL/min
* Hepatitis C with detectable HCV RNA at inclusion
* Positive HBs Ag, except patients with HBeAg-negative chronic HBV infection, previously termed 'inactive carriers' [characterised by the presence of serum antibodies to HBeAg (anti-HBe), undetectable or low (<2,000 IU/mL) HBV DNA levels and normal serum ALT levels] that can be included
* Alcohol intake >210 g/week for men and 140 g/week for women
* Mandatory indication to aspirin or other antiplatelet agents including P2Y12 receptor antagonists according to guidelines of the American Heart Association
* Patient who underwent liver transplantation less than 3 years before screening
* Severe hepatic impairment or significant active liver injury (serum ALT level > 5 times the upper limit of normal values)
* Life expectancy <12 months
* Specific causes of portal hypertension or specific vascular liver diseases: history of bone marrow transplantation, Budd-Chiari syndrome / hepatic venous outflow obstruction, hepatic schistosomiasis diagnosed on liver biopsy (an isolated positive serology is not an exclusion criterion), cardiac failure, Fontan surgery, Abernethy syndrome, Hereditary hemorrhagic telangiectasia, chronic cholestatic diseases, liver infiltration by tumor cells
* Concomitant use of potent inhibitors of CYP3A4 or P-gp. In case of moderate interactions with apixaban (for example, immunosuppressive treatment), the dose of CYP3A4 inhibitor will be adapted according to its plasmatic level in the study patient.
* Hypersensitivity to the active substance or to any of the excipients including lactose.
* Patients unable to give consent (under guardianship or curatorship)
* No written informed consent for participation in the study
* No coverage for medical insurance

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Portal venous system thrombosis | 24 months
  Occurrence or extension of portal venous system thrombosis (including splenic, mesenteric veins, portal trunk or left or right portal branches) at 24 months in patients with INCPH.

SECONDARY OUTCOMES:
Occurrence of side effects | 24 months
  Any major bleeding as defined by the International Society on Thrombosis and Haemostasis guidelines; liver toxicity; adverse events and reactions.
Composite endpoint including thrombosis and major bleeding | 24 months
  Cumulative incidence of one event among: deep vein thrombosis in any location, arterial thrombosis, major bleeding, death
Occurence of vein or arterial thrombosis | 24 months
  Compare the effect of 24 months low dosing of apixaban (2.5 mg x 2/day) versus placebo on one event among: deep vein thrombosis in any location, arterial thrombosis,
Mortality or liver transplantation | 24 months
  cumulative incidence of death (global, liver related, non liver related) or liver transplantation
Complications of liver disease | 24 months
  cumulative incidence of liver decompensation, complications of portal hypertension including portal hypertensive related gastrointestinal bleeding, liver transplantation or death;
Portal hypertension related features | 24 months
  change in size of oesophageal varices
Portal hypertension related features | 24 months
  platelet count
Markers of bacterial translocation and inflammation | 24 months
  circulating concentrations of CRP
Liver function | 24 months
  change in child pugh score
Liver function | 24 months
  change in MELD score
Measure of Quality of life | 24 months
  change in quality of life assessed using SF36 questionnaire
Measure of quality life | 24 months
  change in quality of life assessed using CLDQ questionnaire
occurrence or the extension of portal venous system thrombosis at 24 months after randomisation in patients with INCPH according to HIV status | 24 months
  Compare the effect of 24 months low dosing of apixaban (2.5 mg x 2/day) versus placebo on the occurrence or the extension of portal venous system thrombosis (including splenic, mesenteric veins, portal trunk or left or right portal branches) at 24 months after randomisation in patients with INCPH according to HIV status
predictors of portal venous system thrombosis and liver related events | 24 months
  In group receiving Apixaban : plasma Apixaban levels
predictors of portal venous system thrombosis and liver related events | 24 months
  in the control group : portal blood flow Velocity
predictors of portal venous system thrombosis and liver related events | 24 months
  in the control group : stiffness measured using Fibroscan
predictors of portal venous system thrombosis and liver related events | 24 months
  in the control group : levels of specific coagulation tets (D-dimeres)
treatment compliance | 24 months
  number of compliant patient
occurrence or extension of portal venous system thrombosis or occurrence of deep vein thrombosis in any location or arterial thrombosis in the 6 months after the 24-month treatment with apixaban versus placebo | 30 months
  cumulative incidence of extension of portal venous system thrombosis or deep vein thrombosis in any location or arterial thrombosis in the 6 months after the 24-month treatment with apixaban versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Emmanuel RAUTOU, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Beaujon hospital, Clichy, France, France

IPD SHARING:
Plan to Share IPD: Undecided